CLINICAL TRIAL: NCT01163214
Title: Prospective Randomized Study Comparing Regional Anesthetic Blocks and Periarticular Infiltration for the Management of Postoperative Pain After Total Knee Replacement.
Brief Title: Management of Postoperative Pain After Total Knee Replacement.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mark J. Spangehl, M.D. (Other)
Responsible Party: Sponsor-Investigator, Mark J. Spangehl, M.D., Associate Professor of Orthopedics, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-003312; UL1TR000135 (NIH)
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Results first posted 2014-11-05 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Postoperative Pain; Knee Replacement Arthroplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — Nerve Block; Ropivacaine; Epinephrine; Ketorolac Tromethamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nerve Block (Experimental): Preoperative femoral block with indwelling femoral catheter and a single shot sciatic block.
  Interventions: Drug: Nerve Block
- Periarticular Injection (Active Comparator): Injection combination prior to skin closure.
  Interventions: Drug: Periarticular Injection

INTERVENTIONS:
Drug: Nerve Block — Regional anesthetic nerve block using an indwelling femoral nerve catheter and a single shot sciatic nerve block using 0.5% ropivacaine.
  Other Names: Naropin
  Arms: Nerve Block
Drug: Periarticular Injection — Periarticular local injection into the periarticular soft tissues at the time of knee replacement using a combination of ropivacaine, epinephrine, ketorolac, and morphine sulphate. Subjects in this arm received the injection combination based on three subject weight categories.
  Other Names: Naropin; Adrenalin; Toradol
  Arms: Periarticular Injection

SUMMARY:
The purpose of this study is to compare two methods of postoperative pain management in patients undergoing total knee replacement.

DETAILED DESCRIPTION:
Patients undergoing total knee replacement will be assigned at random to receive one of two methods of postoperative pain management. Patients assigned to nerve block will receive regional anesthetic nerve block using an indwelling femoral nerve catheter and a single shot sciatic nerve block. Patients assigned to periarticular injection will receive periarticular local injection into the periarticular soft tissues at the time of knee replacement using a combination of ropivacaine, epinephrine, ketorolac, and morphine sulphate. Additionally, all patients will be given a standardized combination of oral analgesic medications preoperatively and postoperatively. All patients will receive a posterior stabilized total knee replacement through an medial parapatellar approach.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral primary total knee replacement.
* Weight 50-125 kg.
* Age 18-79 years.
* Intact neurological exam to the surgical lower extremity.
* Cognitively intact with ability to sign informed consent.

Exclusion Criteria:

* Renal insufficiency with creatinine >1.5 mg/dL.
* Allergy to medication used in the study.
* Using narcotic medication prior to surgery (morphine equivalents >=20 mg/day for >7 days.)
* Prior open knee surgery with regional anesthesia or periarticular injection for post-operative pain management.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2010-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Spangehl, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Phoenix, Arizona, United States

REFERENCES:
- [Result] Spangehl MJ, Clarke HD, Hentz JG, Misra L, Blocher JL, Seamans DP. The Chitranjan Ranawat Award: Periarticular injections and femoral & sciatic blocks provide similar pain relief after TKA: a randomized clinical trial. Clin Orthop Relat Res. 2015 Jan;473(1):45-53. doi: 10.1007/s11999-014-3603-0. PMID 24706022

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from Mayo Clinic, Phoenix, Arizona from September 2010 to February 2013.
Period: Overall Study
Arm/Group | Nerve Block | Periarticular Injection
Started | 79 | 81
Completed | 79 | 81
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nerve Block | Periarticular Injection | Total
Number analyzed (Participants) | 79 | 81 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (7.9) | 67.7 (7.2) | 67.7 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 48 | 89
  Male | 38 | 33 | 71
Region of Enrollment [Number; unit: participants]
  United States | 79 | 81 | 160

OUTCOME MEASURES:

1. Secondary Outcome: Pain Scores in the Per-protocol Subset (Participants Who Received the Allocated Treatment)
Description: Pain was measured using a linear analog scale for pain, with a scale from 0 (no pain) to 10 points (worst possible pain).
Time Frame: Afternoon on post-operative Day 1, approximately 14:00
Population: In the nerve block arm 5 subjects were excluded (3 subjects were not treated as planned, and 1 subject received a sciatic catheter instead of a single injection, and 1 subject previously had a nerve block procedure.) In the periarticular injection arm 4 patients were excluded (3 subjects were not treated as planned, and 1 subject was too heavy.)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nerve Block | Periarticular Injection
Number analyzed (Participants) | 74 | 77
units on a scale | 2.9 (2.4) | 3.1 (2.2)
Statistical Analysis 1: Comparison: Nerve Block vs Periarticular Injection; Test type: Superiority or Other; p = 0.78, t-test, 2 sided
Statistical Analysis 2: Comparison: Nerve Block vs Periarticular Injection; Test type: Superiority or Other; p = 0.58, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Post-Operative Pain
Description: as for outcome 1
Time Frame: Afternoon on post-operative Day 1, approximately 14:00
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nerve Block | Periarticular Injection
Number analyzed (Participants) | 79 | 81
units on a scale | 2.9 (2.4) | 3.0 (2.2)
Statistical Analysis 1: Comparison: Nerve Block vs Periarticular Injection; Test type: Superiority or Other; p = 0.76, t-test, 2 sided
Statistical Analysis 2: Comparison: Nerve Block vs Periarticular Injection; Test type: Superiority or Other; p = 0.59, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Narcotic Use
Description: Use of additional narcotic medications (as needed), measured in morphine equivalents.
Time Frame: Intraoperative, Day of surgery, Post-Operative Day 1, Post-Operative Day 2
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Nerve Block | Periarticular Injection
Number analyzed (Participants) | 79 | 81
mg
  Intraoperative | 17.4 (10.1) | 23.6 (8.5)
  Day of Surgery | 4.6 (9.1) | 11.7 (13.1)
  Post-Operative Day 1 | 43.0 (29.0) | 49.0 (29.0)
  Post-Operative Day 2 | 33.0 (28.0) | 30.0 (29.0)
Statistical Analysis 1: Comparison: Nerve Block vs Periarticular Injection; Comparison of arms for intraoperative narcotic use; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Nerve Block vs Periarticular Injection; Comparison of arms for narcotic use on day of surgery as needed; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: Nerve Block vs Periarticular Injection; Comparison of arms for narcotic use on post operative day 1 as needed; Test type: Superiority or Other; p = 0.17, t-test, 2 sided
Statistical Analysis 4: Comparison: Nerve Block vs Periarticular Injection; Comparison of arms for narcotic use on post operative day 2 as needed; Test type: Superiority or Other; p = 0.51, t-test, 2 sided

4. Secondary Outcome: Straight-leg Raise
Description: Post-operative quadriceps function was measured by the number of participants who could perform a straight-leg raise.
Time Frame: Day 1 morning (AM), Day 1 afternoon (PM), Day 2 morning, Day 2 afternoon
Population: The number of participants analyzed varied at each category time point because either data points were missing for participants, or as the condition of the participants improved, they were discharged from the hospital. Number of participants per arm for each time point is shown in each category label.
Measure: Number; unit: participants
Arm/Group | Nerve Block | Periarticular Injection
Number analyzed (Participants) | 78 | 80
participants
  Day 1 AM (Nerve Block=78, Injection=80) | 19 | 63
  Day 1 PM (Nerve Block=76, Injection=78) | 21 | 63
  Day 2 AM (Nerve Block=78, Injection=79) | 52 | 69
  Day 2 PM (Nerve Block=69, Injection=51) | 57 | 42
Statistical Analysis 1: Comparison: Nerve Block vs Periarticular Injection; Comparison between arms for postoperative day 1 morning; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Nerve Block vs Periarticular Injection; Comparison between arms for postoperative day 1 afternoon; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: Nerve Block vs Periarticular Injection; Comparison between arms for postoperative day 2 morning; Test type: Superiority or Other; p = 0.002, t-test, 2 sided
Statistical Analysis 4: Comparison: Nerve Block vs Periarticular Injection; Comparison between arms for postoperative day 2 afternoon; Test type: Superiority or Other; p = 0.97, t-test, 2 sided

5. Secondary Outcome: Length of Stay in Hospital
Description: Length of stay data were calculated from the medical record.
Time Frame: Approximately 2 days after surgery
Population: The number of participants analyzed were different than the baseline values for the arms because data were not available for some participants.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Nerve Block | Periarticular Injection
Number analyzed (Participants) | 74 | 81
days | 2.84 (1.34) | 2.44 (0.65)
Statistical Analysis 1: Comparison: Nerve Block vs Periarticular Injection; Comparison between the arms for length of stay in the hospital; Test type: Superiority or Other; p = 0.02, t-test, 2 sided

6. Secondary Outcome: Number of Subjects Who Experienced Neurological Changes Postoperatively
Description: Participants were questioned at the 6 weeks follow-up visit regarding any neurological changes that were not present preoperatively.
Time Frame: 6 weeks postoperative
Population: The number of participants analyzed in the nerve block arm varied because data were not available for all participants in all neurological categories. The sample size for the periarticular injection arm was 79 because neurological data were not collected on 2 participants.
Measure: Number; unit: participants
Arm/Group | Nerve Block | Periarticular Injection
Number analyzed (Participants) | 78 | 79
participants
  Femoral nerve (nerve block n=77) | 1 | 0
  Common peroneal nerve (nerve block n=78) | 6 | 0
  Tibial nerve (nerve block n=78) | 2 | 1
  Femoral, peroneal, or tibial (nerve block n=77) | 9 | 1
Statistical Analysis 1: Comparison: Nerve Block vs Periarticular Injection; Comparison between arms for femoral nerve; Test type: Superiority or Other; p = 0.49, t-test, 2 sided
Statistical Analysis 2: Comparison: Nerve Block vs Periarticular Injection; Comparison between arms for common peroneal nerve; Test type: Superiority or Other; p = 0.01, t-test, 2 sided
Statistical Analysis 3: Comparison: Nerve Block vs Periarticular Injection; Comparison between arms for tibial nerve; Test type: Superiority or Other; p = 0.62, t-test, 2 sided
Statistical Analysis 4: Comparison: Nerve Block vs Periarticular Injection; Comparison between arms for femoral, peroneal, or tibial nerves; Test type: Superiority or Other; p = 0.009, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected from within 4 days of the surgery.
Arm/Group | Nerve Block | Periarticular Injection
Serious Adverse Events (participants affected / at risk) | 4/79 | 0/81
Other Adverse Events (participants affected / at risk) | 55/79 | 54/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nerve Block (N=79) | Periarticular Injection (N=81)
Acute Pulmonary Embolism (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Lumbar Vertebral Fracture After Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Stroke Middle Cerebral Artery (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nerve Block (N=79) | Periarticular Injection (N=81)
Vomiting (Gastrointestinal disorders) | 19 (19) | 16 (16)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Syncope (Ear and labyrinth disorders) | 3 (3) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 2 (2) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Urinary Retention (Renal and urinary disorders) | 26 (26) | 33 (33)

LIMITATIONS AND CAVEATS:
Participants and staff could not be blinded to the treatment arm received; participants' pain was evaluated at rest and not with activity; the study was not powered to identify certain rare events such as falls.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes